CLINICAL TRIAL: NCT00925236
Title: Phenotypic and Genotypic Identification and Characterization of MYH9-related Constitutional Thrombocytopenia
Acronym: MAGIC-MYH9
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P070110
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: May-Hemalin; Fechtner Syndrome (Disorder); Epstein Syndrome (Disorder); MYH9 Related Disorders
Keywords: MYH9 gene; macrothrombocytopenia; leukocyte inclusions; cataracts deafness; nephritis; MYH9 Related Disorders
MeSH Terms: conditions — MYH9-Related Disorders; Nephritis

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

SUMMARY:
The research involves the establishment of a cohort including as much as possible cases of macrothrombocytopenia related to a "MYH9 syndrome" and the study of mutations and polymorphisms of MYH9 gene in all these patients. As MYH9 syndrome is an autosomal dominant disorder, patients should be heterozygous for a MYH9 gene mutation.

The main goal of our project is looking for correlations between genotype and phenotype. It is planned to characterize the phenotype and genotype of a cohort of patients, including family members that will be addressed during the study in order to better understand the platelet disorder and improve the epidemiological knowledge of MYH9 syndrome. The data will be recorded in a database.

DETAILED DESCRIPTION:
Definition: Extended description of the protocol, including information not already contained in other fields, such as comparison(s) studied. The patients that will participate in the study will be suffering or suspected suffering from MYH9 syndrome.

The study of MYH9 gene will be proposed to the patients but also to both parents of the propositi and other family members (children and adults), whether symptomatic or not. The relatives who will be proved to be heterozygotes for a MYH9 mutation will be considered as new cases and therefore included in the cohort of patients.

Four groups of controls (individuals who are not affected by a decrease in the platelet count) will be constituted:

A1: controls for proplatelets production study A2: controls for platelet proteome study B: controls for MYH9 gene analysis C: controls for leukocytes immunofluorescence study

Patients Patients will be included at the 6 sites of the national Reference Center for Inherited Platelet Disorders (CRPP) after signing an informed consent form. During the visit of inclusion (V1), data usually required for the diagnosis of MYH9 syndrome will be collected: clinical examination, auditory and ocular check, blood tests including MYH9 gene analysis, and search for proteinuria.

Among patients with a MYH9 mutation, a limited number will be recruited in a second step for participating to specific studies focused on the consequences of MYH9 mutations on the proplatelets production and the platelet proteome. The selected patients should be representative of the different phenotypes of MYH9 syndrome. They should be adults and have a platelet count above 50 G / L. A blood sample will be drawn for this purpose during a second visit (V2).

An annual control will be offered at year 1, year 2 and year 3 after inclusion to all the patients confirmed to have MYH9 syndrome (with MYH9 mutation). Each control will include: clinical examination and record of bleeding episodes, if any, during the past year, blood tests, search for proteinuria. The last control (end of the study) will also include auditory and ocular tests.

Relatives The relatives will be included in the study after signing informed consent form during an inclusion visit (VAP) at one of the 6 sites of CRPP. During the visit, a blood sample will be drawn for platelet and MYH9 gene study.

Controls The controls will be included in the study after signing informed consent at 6 sites of the CRPP. During their inclusion visit (VT), a blood sample will be drawn for platelet and MYH9 gene study.

ELIGIBILITY:
Inclusion Criteria:

1. Thrombocytopenia with large/giant platelets (macrothrombocytopenia=MT)
2. and at least one of the following criteria:

   * chronicity of the MT or MT at least found at 2 successive examinations
   * Leukocyte inclusions in polymorphonuclear neutrophils
   * Juvenile sensorineural hearing loss
   * Nephritis
   * Presenile cataracts
   * Familial cases with bleeding disorder associated at least with one of the following symptoms: thrombocytopenia, nephritis, cataracts, deafness, leukocyte inclusions in polymorphonuclear neutrophils
3. Patient who has given his consent
4. Patient who has a social insurance -

Exclusion Criteria:

* Other proven constitutional macrothrombocytopenia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: defined population
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2009-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Study of the correlations phenotype - MYH9 genotype of the patients | final time frame at the end of the study

SECONDARY OUTCOMES:
- Describe the initial clinical symptoms and the long- term evolution of MYH9-related macrothrombocytopenia - Explore the consequences of MYH9 gene mutations on the proplatelets production - Study the effects of MYH9 gene mutations on the platelet | final time frame at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Schlegel, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Robert Debré, Paris, France